CLINICAL TRIAL: NCT04461912
Title: Development of a Medical Device Based on Ultrasounds for Objective Cataract Characterization and Optimal Phacoemulsification Energy Evaluation
Brief Title: Ultrasonic System for Cataract Characterization and Optimal Phacoemulsification Energy Evaluation
Acronym: CATARCTUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Jaime Batista Santos, Investigator Responsible, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: POCI-01-0145-FEDER-028758
Record Dates: First submitted 2020-06-24; First posted 2020-07-08 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Cataract; Ultrasound Therapy; Complications
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: The study includes participants with age-related cataract and healthy subjects as control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cataract (Experimental): Participants with diverse types and severities of cataract, that should realize phacoemulsification surgery
  Interventions: Device: Eye Scan Ultrasound System (ESUS)
- Control (Placebo Comparator): Participants on which the presence of cataract have been excluded
  Interventions: Device: Eye Scan Ultrasound System (ESUS)

INTERVENTIONS:
Device: Eye Scan Ultrasound System (ESUS) — • For the ultrasonic signals acquisitions, an ophthalmic probe working in A-mode scan, must be coupled to the cornea. To reduce the discomfort generated by coupling the probe, topical anaesthesia (oxybuprocaine hydrochloride) will be applied before starting acquisitions. However, if the participant has some known contraindication to this anaesthetic, in replacement, a disposable neutral contact lens will be used as coupling medium between the probe and the cornea.
  The acquisitions are initiated through a starting button in the system's user interface, and the probe must be kept by few seconds for automatic signals records. During this period, signals are visualized in the user interface. Finally the probe is uncoupled, and the acquired signals are saved.

SUMMARY:
This study aims to assess the performance of an ultrasonic system for automatic classification of cataract type and severity, as well as the estimation of the optimal phacoemulsification energy. Ultrasonic signals from the lens will be acquired with the Experimental Medical Device (ESUS) in participants with cataract, and in healthy subjects (control).

The proposed technique may represent an important advance in cataract treatment. The quantitative and automatic classification of cataract type and severity, and the estimation of the optimal phacoemulsification energy is may represent a valuable tool for surgical planning, reducing complications associated to excessive levels of phacoemulsification energy, as well as the times spent on surgeries. This device may be relevant not only for patients, but also for public health systems, reducing waiting lists and associated costs.

DETAILED DESCRIPTION:
This is a prospective, pivotal, non-blinded study. Fifty (50) participants will be recruited at the Coimbra Surgical Center of Portugal. The study will be conducted on subjects with age-related cataract, and on healthy subjects as control group. Since this is a pilot study, no sample size estimation has been implemented. The statistical power will be determined at the end of the study. Only per-protocol participants will be considered on statistical analysis.

Procedures involved. The ultrasonic system (Experimental Medical Device - ESUS) works in A-scan mode, with an acoustic working frequency of 20 MHz. From the ultrasonic signals backscattered from the lenses, acoustic parameters will be extracted, and used for automatic algorithms implementation. This study will be implemented once.

Slit lamp with LOCS III classification will be used as comparator. Contrast sensitivity test results will be used for incipient cataract detection, where slit lamp may present some limitations. Optical coherence tomography and specular microscopy will help on detecting postoperative complications; other complications identified by the physician will be also considered. Surgical parameters as phacoemulsification energy and surgical time will help on phacoemulsification energy evaluation.

Safety assessment. The system uses an ophthalmic probe. There are not anticipated adverse events related to the procedures involved in the use of the ultrasonic system, or any other procedure in the protocol. The safety conditions will be monitored through the occurrence of unanticipated adverse events or serious adverse events. If these situations occur, the event will be reported to the competent authorities (in agreement with the current regulation) and the corrective actions will be implemented.

ELIGIBILITY:
Inclusion criteria:

Cataract group:

* Patients with age-related cataract;
* Indication of phacoemulsification surgery

Control group:

• Patients without cataract

Exclusion criteria:

• Presence of any other ophthalmological condition or systemic disease that could affect the results

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Presence of Cataract | baseline
  Presence of cataract obtained with the Experimental Medical Device (ESUS)

SECONDARY OUTCOMES:
Cataract classification | baseline
  Cataract type and severity obtained with the Experimental Medical Device (ESUS) - based on the LOCS III (Lens Opacity Classification System)
Cataract hardness | before the intervention/procedure/surgery
  Cataract hardness estimated with the Experimental Medical Device (in Gpa)
Phacoemulsification energy | immediately after the intervention/procedure/surgery
  Phacoemulsification energy level estimated with the Experimental Medical Device in the participants performing cataract surgery (considering the phacoemulsification energy parameters provided by the phacoemulsifier).

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Caixinha, PhD, Principal Investigator — miguel.caixinha@gmail.com
Locations (1):
- Centro Cirúrgico de Coimbra (CCCI), Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petrella L, Nunes S, Perdigao F, Gomes M, Santos M, Pinto C, Morgado M, Travassos A, Santos J, Caixinha M. Feasibility assessment of the Eye Scan Ultrasound System for cataract characterization and optimal phacoemulsification energy estimation: protocol for a pilot, nonblinded and monocentre study. Pilot Feasibility Stud. 2022 Sep 29;8(1):219. doi: 10.1186/s40814-022-01173-2. PMID 36175978